CLINICAL TRIAL: NCT04127539
Title: Evaluation of Strong & Steady: A Group Exercise Program for Preventing Functional Decline and Falls Among Community Dwelling Older Adults
Brief Title: Evaluation of Strong & Steady - Fall Preventive Group Exercise Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Glasgow Caledonian University (Other); Fysiofondet (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019/255
Record Dates: First submitted 2019-10-14; First posted 2019-10-15 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Aged
Keywords: Exercise; Fall prevention
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Will start a Strong & Steady group exercise programme immediately after baseline testing.
  Interventions: Behavioral: Strong & Steady exercise program

INTERVENTIONS:
Behavioral: Strong & Steady exercise program — The community-based group exercise program S&S, with strengthening and balance exercise as the main components. The participants will attend a once-weekly, one hour supervised session. The exercises that will be used can be found in the S&S handbook which includes different difficulty levels. All instructors are volunteers and have completed the S&S education. Each exercise session will consist of a warm-up (5-8 min.), endurance exercises (10-15 min.), strength exercises (15 min.), balance exercises (20 min.) and a cool down/stretching (5 min.). In addition to attending the group exercises, the participants will be taught and encouraged to do home exercises twice a week from hand out leaflets that can be found at www.sterkogstodig.no.

SUMMARY:
The aim of the study is to investigate the effect of Strong and Steady (S&S) group exercise on fall risk and physical function among community-dwelling older adults over 12 months. A pre-post test study deign will be used.

DETAILED DESCRIPTION:
The S&S group exercise program builds on the Otago and FaME exercise programs which have shown to be effective in preventing falls. Strong and steady has been adapted to more functionally fit older people.

The study period will be one year. Due to the corona pandemic all S&S groups in Norway have been closed. Due to this all participants have had a break from their exercise program for more than 6 months and can be seen av new participants to the exercise groups. Participants that are about to start in a S&S group in municipalities in Trøndelag will be asked to participate in this study. They will go through tests of muscle strength and balance in addition to questionnaires at baseline and after 6 and 12 months of exercise. Where possible the participants will go through the same tests 1 month before they start to exercise in addition to the three other test timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Able to get to the training facilities on their own
* Able to walk without a walking aid indoors

Exclusion Criteria:

* Diagnosed with dementia

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 95 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
30 sec chair rise | Baseline and 3 months
  Change in number of stands from a chair managed within a time frame of 30 seconds.

SECONDARY OUTCOMES:
Short Physical Performance Battery total score | Baseline, 3, 6 and 12 months
  Includes 5x Sit-to-stand, 4 meters walk test and 3 different 10 sec stance positions. Change in total score (0-12 points).
Number of falls | 12 months
  Number of falls will be collected by daily calendars collected every month
The Short Falls Efficacy Scale-International | Baseline, 3, 6 and 12 months
  The Short Falls Efficacy Scale-International (Short FES-I) questionnaire will be used to assess fear of falling. The total score range from 7 (no concern about falling) to 28 (severe concern about falling). Change in total score will be assessed.
Everyday physical activity | One week monitoring at baseline, 3, 6 and 12 months
  Axivity activity sensors fixed to the lower back ang thigh will be used to measure everyday physical activity. Change in time spent doing physical activity will be assessed.
30 sec chair rise | Baseline, 6 and 12 months
  Change in number of stands from a chair managed within a time frame of 30 seconds.
Four square step test | Baseline, 6 and 12 months
  Time spent doing a sequence of moving through four squares back and fourth.

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn L Helbostad, PhD/Prof, Study Director — The Norwegian University of Science and Technology
Locations (1):
- Norwegian municipalities, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes
Data will be fully anonymised 5 years after study completion and made available for other researcher by request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 5 years after study completion
Access Criteria: By request

REFERENCES:
- See also: The national website for Sterk og stødig — http://sterkogstodig.no